CLINICAL TRIAL: NCT05050123
Title: Comparing a Smartphone-based Virtual Reality Exposure With Standard Relaxation Training for Anxiety on an Inpatient Psychiatric Unit
Brief Title: Smartphone-based Virtual Reality Exposure and Standard Relaxation Training for Anxiety on an Inpatient Psychiatric Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to lack of personnel and budget.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Simon Kung, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-004947
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First episode of anxiety: standard relaxation training (Active Comparator): During a subject's first episode of anxiety the subject will be offered a session of standard relaxation training.
  Interventions: Behavioral: Standard relaxation training
- Second episode of anxiety: virtual reality relaxation (Experimental): During a subject's second episode of anxiety the subject will be offered a session of virtual reality exposure available through the iPhone Google Cardboard virtual reality meditation/relaxation app.
  Interventions: Behavioral: iPhone Google Cardboard virtual reality meditation/relaxation app

INTERVENTIONS:
Behavioral: iPhone Google Cardboard virtual reality meditation/relaxation app — Virtual reality meditation/relaxation app that has 6 scenes of 360° visual imagery with soothing music. The patient can spend about 15 minutes exploring the app.
  Arms: Second episode of anxiety: virtual reality relaxation
Behavioral: Standard relaxation training — 15 minute sessions of guided imagery using Mayo Clinic Patient Education CD-ROM "Relaxation for Your Mind and Body"
  Arms: First episode of anxiety: standard relaxation training

SUMMARY:
The purpose of this study is to compare a smartphone-based virtual reality exposure with standard relaxation training for anxiety and associated symptoms (including pain) on an inpatient psychiatric unit, and whether patients find it usable and beneficial.

DETAILED DESCRIPTION:
The study is open only to inpatients on a specific Mayo Clinic Rochester psychiatric hospital unit, the Mood Disorders Unit. Two different techniques for reducing anxiety will be tried. The first time patients report anxiety, they will be asked to listen to a 15 minute audio CD guiding them through relaxation strategies. The second time patients are anxious, they will be given a cardboard VR goggle set and will view 15 minutes of unguided VR. Before and after each session, they will fill out a short survey of anxiety and related symptoms (including pain ratings) and their reaction to each technique. They will be asked to try each technique at least once during your hospital stay.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized on inpatient Mayo Clinic Mood Disorders psychiatric unit (Generose 3W).

Exclusion Criteria:

* Inability to understand English.
* Patients with primary substance use disorders, primary psychotic disorders, major neurocognitive disorders and active self-harm behaviors and seizure disorders

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, approximately 90 minutes
  Assessment of anxiety with Subjective Units of Distress Scale (SUDS); this 0-100 scale has anchors and guidance for patients to rate their anxiety, 100 is "highest anxiety/distress you have ever felt", 50 is "moderate anxiety/distress; uncomfortable, but can continue to function", and 0 is "no stress; totally relaxed".

SECONDARY OUTCOMES:
Change in associated emotions rating | Baseline, approximately 90 minutes
  The patient will be asked to write up to 3 more associated emotions and rate them 0-10, 10=strongest intensity
Change in pain | Baseline, approximately 90 minutes
  Assessment of pain with Numeric Pain Intensity Scale (NPIS); the scale is measured on a 0-10 scale with 0 equating to no pain and 10 being the most excruciating pain patient has ever felt.
Change in blood pressure | Baseline, approximately 90 minutes
  Measured in mmHg
Change in heart rate | Baseline, approximately 90 minutes
  Measured in beats per minute
Change in respiratory rate | Baseline, approximately 90 minutes
  Measured in breaths per minute

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kung, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials